CLINICAL TRIAL: NCT03004040
Title: Protection From Influenza: Determining the Impact of Prior Infection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Health Sciences North Research Institute (Other)
Collaborators: NOAMA NORTHERN ONTARIO ACADEMIC MEDICINE ASSOCIATION (Unknown)
Responsible Party: Principal Investigator, Janet McElhaney, Vice President of Research and Scientific Director, HSN Volunteer Association Chair in Healthy Aging, Medical Lead for Seniors Care and Consulting Geriatrician, Health Sciences North Research Institute
Other Study IDs: Protection from Influenza
Record Dates: First submitted 2016-12-19; First posted 2016-12-28 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Case: older adult patients (over the age of 65) admitted to Health Sciences North with laboratory confirmed influenza illness (LCII)
  Interventions: Biological: Flu Vaccine
- Control: matched control subjects (non-LCII)
  Interventions: Biological: Flu Vaccine

INTERVENTIONS:
Biological: Flu Vaccine

SUMMARY:
The investigators propose a unique methodology of studying infection and vaccination history and immune responses. As most studies in infection history are conducted on mice, limitations are inherent on their applicability to humans. A longitudinal comparison study following older adults (over the age of 65) hospitalized for influenza are followed through to their hospital discharge and vaccination in the following season. This will allow for the investigation of the course of infection, as well as impact on the response to vaccination.

DETAILED DESCRIPTION:
Significance: This study will provide critical information on the best technique in vaccine candidate testing and improve influenza treatment approaches. The long-term goal of this research is to identify the T-cell responses that are surrogates (biomarkers) of serious complications of influenza in older adults and predict vaccine efficacy (prevention of influenza illness) and vaccine effectiveness (prevention of serious complications). Further, translating new insights into age-related immune dysfunction to the design of new influenza vaccines is critical to addressing this unmet need in the population aged 65 and older.

Innovation: The study will help in the validation of clinical tools and biomarkers as prognostic indicators of influenza illness severity in vaccinated older adults, point-of-care diagnostics that would direct other preventive strategies to reduce the impact of influenza illness in vaccinated older adults, and correlates of protection to evaluate the potential of new influenza vaccines to enhance protection against the serious complications of influenza illness. The investigators have established that GrzB activity and the IFNg: IL-10 ratio in influenza-stimulated PBMC correlate with protection against influenza, and preliminary data to show that low GrzB activity in influenza-stimulated PBMC correlates with more severe disease and higher levels of frailty. The innovations of this project are the established methods for developing correlates of protection, the clinical insights into how frailty affects immune-mediated protection against influenza, and the direct translation of this research to provide a reasonable method for primary care clinicians to estimate vaccine effectiveness in an individual older person. These results will translate to the practical design of clinical trials to evaluate the potential for new influenza vaccines to better protect against the serious complications of influenza and complement those based on antibody titers and/or clinical outcomes alone.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent provided by the participant.
2. Age 65 years of age or older admitted to Health Sciences North with at least one the following:

   * Laboratory confirmed influenza illness
   * Acute exacerbation of chronic obstructive pulmonary disease (AECOPD).
   * Any respiratory or influenza-like symptoms (dyspnea, cough, sore throat, myalgia, arthralgia, fever, delirium/altered level of consciousness) that a test for influenza was negative.
3. Willing to receive influenza vaccination in the subsequent flu season

Exclusion Criteria:

1. Patients whose reason for hospital admission was unrelated to influenza or (for example patients admitted due to trauma, elective surgery, or patients who have an alternative diagnosis that is clearly not respiratory).
2. Chest x-ray positive for pneumonia.
3. Study participants who cannot be vaccinated due to previous severe reaction to influenza vaccine, egg, latex, or thimerosol allergies, or refusal of vaccination.
4. Immunosuppressive disorders or medications (including oral prednisone in doses >10 mg daily).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Older adult patients (over the age of 65) admitted to Health Sciences North with laboratory confirmed influenza illness (LCII) and matched control subjects (non-LCII).
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-12; Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
High expression of CTL associated cytokines and granzymes in PBMC's are predictors of influenza infection severity. | 2 years
  PBMCs from adults hospitalized for laboratory confirmed influenza illness (LCII) will be collected at admission and 30 days post hospitalization. These samples will be matched with hospitalized non-LCII adult controls. T-cells will be isolated from whole blood samples and gene expression of IFNg, IL10 and GrzB will be measured and compared between time points and subjects. These levels do not have a separate unit of measure.

SECONDARY OUTCOMES:
Vaccination in previously infected individuals increases the protection provided by subsequent vaccination and will be higher than those receiving vaccination alone (with no previous infection) | 2 years
  Older adults hospitalized for influenza illness the previous season will be compared to matched, hospitalized older adults with influenza-like illness (non-LCII). PBMCs will be collected from each group, before receiving influenza vaccination and 4 weeks after vaccination. PBMCs will be challenged ex vivo with influenza virus and gene expression of CTL related genes will be measured and compared between each group.

CONTACTS AND LOCATIONS:
Locations (1):
- Health Sciences North Research Institute, Greater Sudbury, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No